CLINICAL TRIAL: NCT04165694
Title: Single Anastomosis Duodenal Ileal Bypass (SADI) as a Second Stage for Sleeve Gastrectomy Weight Loss Failure
Brief Title: Single Anastomosis Duodenal Ileal Bypass (SADI) for Sleeve Revision
Acronym: SADI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12208
Record Dates: First submitted 2019-11-07; First posted 2019-11-18 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Bariatric Surgery Candidate; Severe Obesity
Keywords: weight loss failure; laparoscopic sleeve gastrectomy
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: The study is a pre-/post-test prospective intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Single Anastomosis Duodenal Ileal Bypass (SADI) — The purpose of the research is to study additional weight loss and resolution of comorbidities in patients who undergo revision of their sleeve gastrectomy to a Single Anastomosis Duodenal Ileal bypass (SADI). The sleeve gastrectomy which you have already undergone is now the most common bariatric procedure performed. This operation was part of a 2-stage operation known a Duodenal Switch (DS) which was a sleeve gastrectomy followed by a long bypass of the intestine that involved 2 connections. This operation has many complications such as vitamin deficiencies and potential malnutrition. The SADI procedure is a version of the DS that bypasses less of the intestine and one less connection of the small bowel.

SUMMARY:
The goal of this study is two part: 1) to add to the literature which is still somewhat sparse with numbers of patients undergoing the Single Anastomosis Duodenal Ileal Bypass (SADI) as a revision for laparoscopic sleeve gastrectomy (LSG) and 2) to have a treatment option for our Kaiser Permanente patients who seek additional assistance after a LSG with persistent morbid obesity and the comorbidities that come with it.

DETAILED DESCRIPTION:
Patients will be recruited during 10/15/2019 through 12/31/2022 with the following inclusion criteria: 1) body mass index (BMI) 35 - 39 kg/m2 with comorbid conditions; 2) BMI 40+ kg/m2 with no comorbidities; 3) having a previous LGS; 4) having lost less than 10% total weight loss with this LSG; 5) being a Kaiser member at the time of surgery; and 6) being at least 18 years of age. Exclusion criteria will include: 1) BMI less than 35; 2) having a hiatal hernia; 3) having severe Gastroesophageal Reflux Disease; 4) having a primary bariatric procedure other than LSG; 5) having already had a revisional bariatric procedure; and 6) being less than 18 years old.

Age range for participants will be 18 - 100 years old. We will recruit 50 patients.

Revisional procedures for weight regain are PART OF USUAL CARE at Kaiser Permanente Southern California. However SADI is a type of revisional procedure that is still considered experimental. This procedure has a single surgical anastomosis. It has a restrictive component when reducing the greater curvature of the stomach, but specially a malabsorptive component, as the common channel is also reduced. The objective of this surgical technique is to lessen the intestinal loop where nutrients are absorbed. It was part of a more extreme procedure, that is currently standard of care, called the Duodenal Switch (DS).

The DS procedure which is PART OF USUAL CARE results in very successful massive weight loss however, it also has severe complications especially vitamin deficiencies.

The SADI procedure is thought to confer the same weight loss benefits of the DS but without the severe complications. This has not been tested systematically.

These eligibility criteria will be verified by the bariatric surgeon who is doing the consult for a revisional procedure AS PART OF USUAL CARE. This will entail the surgeon looking in the electronic medical record before meeting with the patient.

However, this review of the medical record before surgical consult is PART OF USUAL CARE.

All data collection and study follow-up visits are PART OF USUAL CARE for bariatric patients at Kaiser Permanente Southern California. THIS INCLUDES PATIENTS WHO RECEIVE REVISIONAL SURGERY. The only part of the study that is not usual care is the surgical procedure itself. The patients enrolled in the proposed study will receive the following visits AS PART OF USUAL CARE:

1. Surgical consult 2 - 6 weeks before surgery at which point the patients will be offered the SADI procedure and consent will be done by the surgeon doing the consult in person in the surgeon's office in the Department of Surgery at the West Los Angeles Medical Center.
2. Visit with bariatric physician 7 - 10 days before surgery to go over laboratory values and to insure instructions for surgical preparation were followed.
3. Visit with surgeon and bariatric physician 7 - 10 days after surgery.
4. Visit with bariatric physician 4 - 6 weeks after surgery.
5. Visit 6 months after surgery with surgeon, bariatric physician, and other te am members as necessary (i.e. nutritionist or social worker).
6. Visit 12 months after surgery with surgeon, bariatric physician, and other team members as necessary (i.e. nutritionist or social worker).
7. Annual phone calls at years 1, 2 and 3 after surgery with bariatric care manager to monitor laboratory measures, weight loss, and complications.

All data to evaluate the effectiveness of SADI will be abstracted from the electronic medical record, These measures are taken from the patients as PART OF US UAL CARE. There are no specific measures added to usual care for the SADI procedure. We already have a protocol for the DS procedure. These data will include weight, height, laboratory results, diagnoses, utiliza tion of services, and pharmacy records. No questionnaires will be used in this study.

For each patient, data will be abstracted for 12 months before surgery and up to 3 years after surgery. No questionnaires will be administered.

The primary outcome for the study will be percent total weight loss at 3 years calculated as (weight at surgery - weight at 3 years)/weight at surgery. Data will be analyzed using linear regression to predict what factors at baseline such as disease burden, gender, age, race ethnicity, and BMI predict percent total weight loss at 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Body Mass Index (BMI) 35 - 39 kg/m2 with comorbid conditions; OR
2. BMI 40+ kg/m2 with no comorbidities; AND
3. having a previous laparoscopic sleeve gastrectomy (LGS); AND
4. having lost less than 10% total weight loss with this LSG; AND
5. being a Kaiser member at the time of surgery; AND
6. being at least 18 years of age.

Exclusion Criteria:

1. BMI less than 35 kg/m2; OR
2. having a hiatal hernia; OR
3. having severe Gastroesophageal Reflux Disease; OR
4. having a primary bariatric procedure other than LSG; OR
5. having already had a revisional bariatric procedure; OR
6. being less than 18 years old.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent Total Weight Loss (change in weight relative to baseline) | 3 years
  This is weight loss relative to the initial body weight at the time of surgery calculated as (weight at surgery - weight at follow-up)/weight at surgery. This is already a change score.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Southern California West Los Angeles Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No